CLINICAL TRIAL: NCT02579096
Title: CSP #594 - Comparative Effectiveness in Gout: Allopurinol vs. Febuxostat
Brief Title: CSP594 Comparative Effectiveness in Gout: Allopurinol vs. Febuxostat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 594
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Gout; Chronic Kidney Diseases
Keywords: Gout; Allopurinol; Febuxostat; CKD
MeSH Terms: conditions — Gout; Renal Insufficiency, Chronic | interventions — Allopurinol; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allopurinol / Sham Comparator (Febuxostat) (Active Comparator): Patients will be titrated up to the dose that will lower to target uric acid levels. A placebo resembling Febuxostat will be given with allopurinol
  Interventions: Drug: allopurinol capsule, 100-800 mg by mouth once daily; Drug: Placebo, vehicle control (febuxostat-shaped)
- Febuxostat / Sham Comparator (Allopurinol) (Active Comparator): Febuxostat will be titrated up to the dose that will lower to target uric acid levels. A placebo resembling Allopurinol will be given with Febuxostat
  Interventions: Drug: febuxostat tablet 40-120 mg by mouth once daily; Drug: Placebo, vehicle control (allopurinol-shaped)

INTERVENTIONS:
Drug: allopurinol capsule, 100-800 mg by mouth once daily — Patients will be up-titrated up to the dose required to reach target uric acid levels.
  Other Names: Zyloprim; CAS: 315-30-0
  Arms: Allopurinol / Sham Comparator (Febuxostat)
Drug: febuxostat tablet 40-120 mg by mouth once daily — Patients will be up-titrated to the dose required to reach target uric acid levels.
  Other Names: Uloric; CAS: 144060-53-7; NDCs: 64764-677-11, 64764-677-13, 64764-677-19, 64764-677-30, 64764-918-11, 64764-918-18, 64764-918-30, 64764-918-90
  Arms: Febuxostat / Sham Comparator (Allopurinol)
Drug: Placebo, vehicle control (febuxostat-shaped) — Placebo tablets resembling febuxostat will be given with allopurinol.
  Arms: Allopurinol / Sham Comparator (Febuxostat)
Drug: Placebo, vehicle control (allopurinol-shaped) — Placebo capsules resembling allopurinol will be given with febuxostat.
  Arms: Febuxostat / Sham Comparator (Allopurinol)

SUMMARY:
This trial will compare two effective therapies, allopurinol and febuxostat, to lower serum uric acid and therefore prevent further gout attacks. These therapies have never been compared at appropriate doses. Further, they will be studied in patients with kidney disease for the first time.

DETAILED DESCRIPTION:
Gout is the most common form of inflammatory arthritis affecting adults (1), with a disease frequency that continues to increase dramatically (2). Gout is associated with substantial morbidity and mortality which are concentrated in older men and magnified in patients with chronic kidney disease (CKD) (3-6), demographics common to the Veterans Affairs (VA) Health System. Effective gout therapies are readily available and are centered primarily on the use of approved urate lowering therapy (ULT). Despite having excellent ULT options available to patients (7), gout is extremely poorly managed especially in patients with CKD (8-10).

The two most widely used ULTs in clinical practice, allopurinol and febuxostat, have recently been endorsed as the two acceptable first-line treatment strategies in chronic gout (7). Although both agents appear to be efficacious and generally well-tolerated, allopurinol and febuxostat have significantly different costs and have never been compared to each other at appropriate doses. Randomized controlled trials completed to date comparing allopurinol with febuxostat in gout have used 'fixed' and, in many cases, insufficient doses of allopurinol (11-13), an approach that is contrary to current guideline recommendations (7). Furthermore, these studies have included only very small proportions of gout patients with CKD even though CKD is present in approximately 1 of every 2 gout sufferers (14).

To test the hypothesis that allopurinol is non-inferior to febuxostat in the treatment of gout, the investigators propose a randomized open-label non-inferiority trial, which for the first time compares allopurinol with febuxostat using appropriately titrated doses and a "treat-to-target" approach. Further, the investigators will assess the comparative effectiveness of these agents in a significant number of gout patients with co-morbid CKD.

The investigators plan to enroll 950 participants with a diagnosis of gout, including participants with stage 3 CKD, who are hyperuricemic defined as a serum uric acid concentration (sUA) above 6.8 mg/dl. Participants will be recruited from 18 Veteran Affairs and 5 Rheumatology and Arthritis Investigational Network (RAIN) sites. The total duration of the trial will be 4 years. Recruitment will occur over 24 months. Participants will be followed for 72 weeks. This will include a 24 week Dose Titration Phase (Phase 1) followed by a 24 week Maintenance and Optimization Phase (Phase 2) and then a 24 week Steady State Flare Observation Phase (Phase 3). The investigators will use a "treat-to-target" approach with specified titration of ULT dosing to obtain goal sUA. Maximal daily drug doses will be 800 mg/day for allopurinol or 120 mg/day for febuxostat.

The primary outcome will be the proportion of participants who have at least one gout flare in the allopurinol group compared to the febuxostat group during Phase 3. This primary outcome was endorsed by the patient and VA provider groups that were surveyed (see below). All participants will be followed during Phase 3 regardless of the achievement of sUA goal. The primary hypothesis will test the non-inferiority of allopurinol with regards to proportions of flares. The investigators anticipate that approximately 15 to 20% of patients will flare during Phase 3.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* History of gout - crystal proven or historical as defined by ACR criteria listed above
* Serum urate level > 6.8 mg/dl

Exclusion Criteria:

* Stage 4 or 5 Chronic Kidney Disease (CKD) - defined as eGFR < 30 ml/min/1.73 m2
* Women less than 50 years of age
* Patients with a history of prior solid organ / hematopoietic transplantation
* Previous allergy or intolerance to allopurinol or febuxostat
* Patients who are not candidates for any of the recommended prophylactic medications (colchicine, naprosyn or glucocorticoids)
* Patients who in the opinion of the investigator have a high genetic risk for allopurinol hypersensitivity syndrome (AHS*) unless they have been found to be negative for HLA B5801.
* Previous history of failure to reach target uric acid levels despite therapy with allopurinol at dose > 300 mg/day
* Prior febuxostat use
* Patients with malignancies that are currently active with exception of non-melanoma skin cancer
* Patients with serum uric acid levels >15 mg/dl
* Patients with myelodysplasia and hemoglobin of < 8.5 mg/dL
* Patients with chronic liver disease with more than one of the following:

  * INR > 1.7, not on Warfarin therapy
  * Bilirubin 2 mg/dL
  * Serum albumin < 3.5 mg/dL
  * Ascites
  * Encephalopathy
* Current use of azathioprine, mercaptopurine, didanosine, cyclophosphamide, probenecid, lesinurad or pegloticase
* Enrollment in another randomized interventional clinical trial
* Any severe medical condition that, in the enrolleer's opinion, is likely to compromise the participant's ability to complete the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R O'Dell, Study Chair — Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE
Locations (23):
- United States (23):
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Mayo Clinic Rochester MN ? RAIN 1, Rochester, Minnesota
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - University of Nebraska Medical Center ? RAIN 5, Omaha, Nebraska
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Sanford Bismarck Medical Center ? RAIN 2, Bismarck, North Dakota
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Yankton Medical Clinic ? RAIN 3, Yankton, South Dakota
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont
  - Salem VA Medical Center, Salem, VA, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be made available after study closure only to research credentialed Veterans Affairs researchers who submit a valid study question to their IRB of record. A Data Use Agreement will be in effect between the researcher and the coordinating center
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After primary and secondary analyses and subsequent publications
Access Criteria: Executed data use agreement with CSP Coordinating Center approval
URL: https://www.research.va.gov/programs/csp/default.cfm

REFERENCES:
- [Background] Timilsina S, Brittan K, O'Dell JR, Brophy M, Davis-Karim A, Henrie AM, Neogi T, Newcomb J, Palevsky PM, Pillinger MH, Pittman D, Taylor TH, Wu H, Mikuls TR. Design and Rationale for the Veterans Affairs "Cooperative Study Program 594 Comparative Effectiveness in Gout: Allopurinol vs. Febuxostat" Trial. Contemp Clin Trials. 2018 May;68:102-108. doi: 10.1016/j.cct.2018.03.015. Epub 2018 Mar 27. PMID 29597007
- [Result] O'Dell JR, Brophy MT, Pillinger MH, Neogi T, Palevsky PM, Wu H, Davis-Karim A, Newcomb JA, Ferguson R, Pittman D, Cannon GW, Taylor T, Terkeltaub R, Cannella AC, England BR, Helget LN, Mikuls TR. Comparative Effectiveness of Allopurinol and Febuxostat in Gout Management. NEJM Evid. 2022 Mar;1(3):10.1056/evidoa2100028. doi: 10.1056/evidoa2100028. Epub 2022 Feb 3. PMID 35434725
- [Derived] Sanchez C, Campeau A, Liu-Bryan R, Mikuls TR, O'Dell JR, Gonzalez DJ, Terkeltaub R. Effective xanthine oxidase inhibitor urate lowering therapy in gout is linked to an emergent serum protein interactome of complement and inflammation modulators. Sci Rep. 2024 Oct 19;14(1):24598. doi: 10.1038/s41598-024-74154-5. PMID 39426967
- [Derived] Sanchez C, Campeau A, Liu-Bryan R, Mikuls TR, O'Dell JR, Gonzalez DJ, Terkeltaub R. Effective xanthine oxidase inhibitor urate lowering therapy in gout is linked to an emergent serum protein interactome of complement activation and inflammation modulators. Res Sq [Preprint]. 2024 May 9:rs.3.rs-4278877. doi: 10.21203/rs.3.rs-4278877/v1. PMID 38766125
- [Derived] Sanchez C, Campeau A, Liu-Bryan R, Mikuls T, O'Dell J, Gonzalez D, Terkeltaub R. Sustained xanthine oxidase inhibitor treat to target urate lowering therapy rewires a tight inflammation serum protein interactome. Res Sq [Preprint]. 2024 Jan 2:rs.3.rs-3770277. doi: 10.21203/rs.3.rs-3770277/v1. PMID 38260556

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 950 subjects were enrolled into the study. However, 10 subjects were excluded from study participation :
  * 3 due to screening errors
  * 7 dropped out before receiving study treatment
Groups:
- Allopurinol / Sham Comparator (Febuxostat): Patients will be up-titrated up to the dose required to reach target uric acid levels.
  Allopurinol: allopurinol capsule, 100-800 mg by mouth once daily
  Placebo: tablets resembling febuxostat will be given with allopurinol.
- Febuxostat / Sham Comparator (Allopurinol): Patients will be up-titrated to the dose required to reach target uric acid levels.
  Febuxostat: tablet 40-120 mg by mouth once daily
  Placebo: capsules resembling allopurinol will be given with febuxostat.
Period: Phase 1, Weeks 0 - 24
Arm/Group | Allopurinol / Sham Comparator (Febuxostat) | Febuxostat / Sham Comparator (Allopurinol)
Started | 468 | 472
Completed | 411 | 422
Not Completed | 57 | 50
Not completed — Side effects with study medications | 10 | 6
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 32 | 36
Not completed — Lost to Follow-up | 9 | 4
Not completed — Other reasons | 4 | 3
Period: Phase 2, Weeks 25 - 48
Arm/Group | Allopurinol / Sham Comparator (Febuxostat) | Febuxostat / Sham Comparator (Allopurinol)
Started | 411 | 422
Completed | 389 | 391
Not Completed | 22 | 31
Not completed — Death | 2 | 4
Not completed — Side effects with study medications | 3 | 1
Not completed — Physician Decision | 4 | 0
Not completed — Withdrawal by Subject | 9 | 12
Not completed — Lost to Follow-up | 4 | 9
Not completed — Other reasons | 0 | 5
Period: Phase 3, Weeks 49 - 72
Arm/Group | Allopurinol / Sham Comparator (Febuxostat) | Febuxostat / Sham Comparator (Allopurinol)
Started | 389 | 391
Completed | 367 | 373
Not Completed | 22 | 18
Not completed — Death | 3 | 2
Not completed — Side effects with study medications | 0 | 1
Not completed — Physician Decision | 0 | 5
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Lost to Follow-up | 10 | 5
Not completed — Participant required to take exclusion medication on a regular basis | 0 | 1
Not completed — Other reasons | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Allopurinol / Sham Comparator (Febuxostat): Patients will be titrated up to the dose that will lower to target uric acid levels. A placebo resembling febuxostat will be given with allopurinol
  allopurinol: Patients will be titrated up to the dose that will lower to target uric acid levels.
  Placebo, vehicle control (febuxostat-shaped): Placebo in the shape of febuxostat will be given with allopurinol
- Febuxostat / Sham Comparator (Allopurinol): febuxostat will be titrated up to the dose that will lower to target uric acid levels. A placebo resembling Allopurinol will be given with febuxostat
  febuxostat: febuxostat will be titrated up to the dose that will lower to target uric acid levels.
  Placebo, vehicle control (allopurinol-shaped): Placebo in the shape of allopurinol will be given with febuxostat
- Total: Total of all reporting groups
Arm/Group | Allopurinol / Sham Comparator (Febuxostat) | Febuxostat / Sham Comparator (Allopurinol) | Total
Number analyzed (Participants) | 468 | 472 | 940
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (11.8) | 61.3 (12.9) | 62.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 461 | 464 | 925
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 27 | 47
  Not Hispanic or Latino | 444 | 443 | 887
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 14 | 15 | 29
  Native Hawaiian or Other Pacific Islander | 10 | 9 | 19
  Black or African American | 104 | 102 | 206
  White | 315 | 322 | 637
  More than one race | 10 | 7 | 17
  Unknown or Not Reported | 12 | 15 | 27
CKD3 [Count of Participants; unit: Participants] — Participants with Chronic kidney disease stage 3 (CKD3). CKD3 is defined as having eGFR = 30-59 mL/min/1.73m^2
  Participants | 181 | 170 | 351
Tophus [Count of Participants; unit: Participants] — Participants with tophus
  Participants | 81 | 71 | 152
sUA >= 9 mg/dL [Count of Participants; unit: Participants] — Participants with Serum Uric Acid (sUA) >= 9 mg/dL
  Participants | 160 | 148 | 308
Pre-study allopurinol users with dose <= 300 mg [Count of Participants; unit: Participants] | 178 | 167 | 345

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing ≥ 1 Gout Flare During Phase 3
Description: Participants were defined as flaring in Phase 3 if they:
  -1) met 3 of 4 following participant-reported criteria:
  * a) warm joint(s)
  * b) swollen joint(s)
  * c) pain (>3) at rest on a scale of 0-10 (10 being the worst pain)
  * d) self-identified gout flare
  OR
  -2) reported use of medications to treat flare
Time Frame: Phase III of the study (weeks 49-72 of study duration)
Population: Primary analysis excluded patients who either never received the trial interventions, or were identified as ineligible after randomization, or dropouts; a complete case analysis was conducted on total of 749 subjects: 740 who completed phase 3 of the study plus 9 subjects who terminated in phase 3 after having an outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Allopurinol / Sham Comparator (Febuxostat) | Febuxostat / Sham Comparator (Allopurinol)
Number analyzed (Participants) | 370 | 379
Participants | 135 | 165
Statistical Analysis 1: Comparison: Allopurinol / Sham Comparator (Febuxostat) vs Febuxostat / Sham Comparator (Allopurinol); One-sided null hypothesis posited that allopurinol was inferior to febuxostat. The proportions of participants with ≥ 1 gout flare during phase 3 were compared between the two treatments; Test type: Non-Inferiority — A non-inferiority bound of 8% was established during the trial design; a one-sided alpha level was set at 0.05; p < 0.001, t-test, 1 sided; Risk Difference (RD) = -7, 95% CI 1-sided [upper limit -1.2]

ADVERSE EVENTS:
Time Frame: Beginning at informed consent and continuing until the end of participation in the study at 72 weeks, plus 30 days of observation.
Description: Data on adverse events was collected spontaneously through patient reports, actively elicited during visits through open-ended questioning and examination, and gathered at the time of telephone contact and medical record reviews during the follow-up period.
Arm/Group | Allopurinol / Sham Comparator (Febuxostat) | Febuxostat / Sham Comparator (Allopurinol)
All-Cause Mortality (participants affected / at risk) | 8/468 | 8/472
Serious Adverse Events (participants affected / at risk) | 125/468 | 123/472
Other Adverse Events (participants affected / at risk) | 36/468 | 44/472
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopurinol / Sham Comparator (Febuxostat) (N=468) | Febuxostat / Sham Comparator (Allopurinol) (N=472)
Anaemia (Blood and lymphatic system disorders) | 2 (5) | 3 (5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 4 (4) | 3 (4)
Arrhythmia supraventricular (Cardiac disorders) | 12 (18) | 8 (11)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 27 (56) | 12 (19)
Coronary artery disease (Cardiac disorders) | 3 (3) | 2 (2)
Hypertensive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4) | 8 (8)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (3)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 5 (5) | 4 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 5 (5) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acute haemorrhagic conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 6 (6) | 12 (15)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 3 (3)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 2 (2)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (4) | 3 (3)
Pneumonia (Infections and infestations) | 10 (11) | 9 (10)
Postoperative wound infection (Infections and infestations) | 3 (3) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 6 (8)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 7 (8)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Gout (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 7 (7)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 3 (3)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
IIIrd nerve paresis (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 2 (2) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Substance use disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (5) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 19 (24) | 12 (12)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Alcohol detoxification (Surgical and medical procedures) | 1 (1) | 0 (0)
Aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 2 (2) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 2 (2) | 2 (2)
Knee arthroplasty (Surgical and medical procedures) | 2 (2) | 4 (4)
Lung lobectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Metabolic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Pancreaticosplenectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Prostatic operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal operation (Surgical and medical procedures) | 0 (0) | 2 (2)
Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Tenoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopurinol / Sham Comparator (Febuxostat) (N=468) | Febuxostat / Sham Comparator (Allopurinol) (N=472)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 8 (9)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (7)
Alanine aminotransferase increased (Investigations) | 18 (18) | 21 (22)
Drug eruption (Skin and subcutaneous tissue disorders) | 11 (11) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT02579096/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT02579096/SAP_002.pdf
  • Informed Consent Form (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT02579096/ICF_000.pdf